CLINICAL TRIAL: NCT00013793
Title: Ultrasound and Motivational Enhancement for Prenatal Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NCRR-M01RR02558-0153
Record Dates: First submitted 2001-03-29; First posted 2001-03-30 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Pregnancy; Smoking
MeSH Terms: conditions — Smoking | interventions — High-Energy Shock Waves

INTERVENTIONS:
Behavioral: Motivational enhancement and ultrasound

SUMMARY:
The primary purpose of this randomized clinical trial is to test the efficacy of motivational enhancement (ME) therapy combined with biologic feedback (fetal ultrasound) for increasing smoking quit rates among low-income pregnant women considered resistant smokers. We hypothesize that ME along with biofeedback will increase the rate of validated smoking cessation at 8 months gestation by at least 10 percentage points above that produced by "Best Practice" (BP) counseling alone. This study will also examine reduction of smoking among non-quitters and maintenance of smoking cessation through 6 weeks postpartum among women who quit.

Prenatal smoking is the leading preventable cause of low birth weight in the US. Reduction in smoking during pregnancy could result in significant improvements in pregnancy outcomes and reducing the cost of health care. There is evidence that low-intensity pregnancy smoking cessation programs may be inadequate for women who are more addicted, and at educational and economic disadvantage. Motivational enhancement strategies have shown considerable promise in the treatment of addictive behaviors. Physiological feedback highlighting prenatal effects of smoking and benefits of cessation has been found to enhance prenatal smoking cessation counseling. An intervention that combines motivational enhancement counseling and physiological feedback may have powerful effects beyond low-intensity interventions or usual counseling.

DETAILED DESCRIPTION:
Targeting women who deliver at one of the two UT-Houston teaching hospitals, Lyndon B. Johnson (LBJ) and Hermann Hospitals, pregnant women between 18 and 28 weeks gestation will be recruited from University of Texas/Harris County Hospital District-affiliated clinics, including Acres Homes, Aldine, Settegast, Baytown, and Squatty Lyons, LBJ and Hermann Hospital outpatient clinics, private practice OB/GYN's with patients who will deliver at Hermann Hospital, and area WIC (Women, Infants and Children) Program sites. Participants will be randomized to one of three groups, including 1) best practice (BP) counseling, 2) BP plus ultrasound, and 3) BP plus ultrasound plus motivational enhancement (ME) counseling. Counseling and cotinine testing will be performed at the University Clinical Research Center (UCRC) initially, at 34 weeks, and at 6 weeks postpartum. The primary outcome is the rate of smoking cessation among the women at 34 weeks gestation. Based on previous reports, projected quit rates for the 3 interventions, BP, BP + ultrasound, and BP + ultrasound + ME are .06, .12, and .20, respectively. A sample size of 360 will be necessary in order to observe these differences in quit rates. The chi-square test for trend in proportions will be used to determine statistical significance for this primary outcome.

ELIGIBILITY:
Inclusion Criteria: Pregnant women who are smokers, 16 years and older, 15-28 weeks gestation

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Janet Y. Groff, M.D., Ph.D., Principal Investigator
Locations (1):
- University of Texas Medical School, Houston, Texas, United States